CLINICAL TRIAL: NCT02737293
Title: Whole Egg Intake and the Mediterranean Diet
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 and expiration of grant funds
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GFHNRC147
Record Dates: First submitted 2016-03-31; First posted 2016-04-13 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Diet (Experimental): Menu based on the average American diet.
  Interventions: Other: Control Diet
- Med Diet (Experimental): Menu based on the typical Mediterranean diet (Med Diet) pattern.
  Interventions: Other: Med Diet
- Med Diet + Whole Egg (Experimental): Menu based on the typical Mediterranean diet (Med Diet) pattern with the addition of 1 whole egg per 1000 kilocalories.
  Interventions: Other: Med Diet + Whole Egg

INTERVENTIONS:
Other: Control Diet — 4-week intake of Control Diet 5 day rotating menu
  Arms: Control Diet
Other: Med Diet — 4-week intake of Med Diet 5 day rotating menu
  Arms: Med Diet
Other: Med Diet + Whole Egg — 4-week intake of Med Diet plus Whole Egg 5 day rotating menu
  Arms: Med Diet + Whole Egg

SUMMARY:
This project will evaluate the daily intake of whole eggs in the Mediterranean Diet (Med Diet). Cholesterol levels are normally related to cardiovascular disease (CVD) risk. Dietary fat and the total diet makeup are well known modifiers of CVD risk. The Med Diet has been shown to decrease blood lipids (fats) and reduce inflammation. Cholesterol intake from eggs may not be as bad as once thought and, in fact, may help to improve the blood lipid (fat) levels. This study is being done to test how the addition of eggs to a Med Diet affects blood lipids and other risk markers for CVD.

DETAILED DESCRIPTION:
Elevated serum cholesterol is a major contributor to cardiovascular disease (CVD), which is responsible for ~1/3 of all deaths in the US. However, about 50% of those who experience heart attacks have normal cholesterol levels. Cholesterol is carried in lipoproteins (HDL, LDL, and VLDL) and the amount in circulation is used to evaluate CVD risk. However, the particle size and density of lipoprotein subfractions may be more predictive for atherogenesis than their total levels. Dietary fatty acids are well recognized modulators of lipoproteins, and ultimately CVD risk. Saturated and trans fatty acids have a negative effect on CVD risk while poly- and monounsaturated fatty acids (PUFA, MUFA) appear to be protective. The Mediterranean Diet (Med Diet) decreases atherogenic lipoproteins and reduces systemic inflammation. It is unknown how high cholesterol intake within a Med Diet will affect these parameters, although recent evidence implies that the fatty acid content of the diet is more important than the cholesterol content. Therefore, this project will evaluate the daily inclusion of whole eggs, a high cholesterol food, in the Med Diet on lipid profiles, lipoprotein particle size and density and biomarkers of systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with the demands of the experimental protocol
* Not performing vigorous exercise >2 times per week
* BMI 25-39.9 kg/m2
* Non-nicotine-using

Exclusion Criteria:

* Have an egg allergy
* Have diabetes
* Have high triglyceride levels
* Have uncontrolled high blood pressure
* Have used tobacco products or nicotine in any form including snuff, pills and patches, or e-cigarettes in the previous 6 months
* Use prescription medications or over-the-counter lipid lowering drugs (such as statins) or anti-inflammatory medications (such as aspirin, ibuprofen or Aleve) on a regular basis
* Take omega 3 supplements, plant sterols or sterol esters
* Are pregnant or lactating
* Have been diagnosed with an eating disorder
* Inability to give consent
* Unwillingness or inability to consume the treatment diets

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Change in lipoprotein metabolism | baseline and 4 weeks
  Assess lipid metabolism response to the intervention.

SECONDARY OUTCOMES:
Change in inflammatory markers | baseline and 4 weeks
  Determine inflammatory marker response to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Picklo, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT02737293/ICF_000.pdf